CLINICAL TRIAL: NCT00505427
Title: Alpha Lipoic Acid and Polycystic Ovary Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8476-27691-01
Record Dates: First submitted 2007-07-20; First posted 2007-07-23 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2013-06

CONDITIONS: Insulin Resistance; Oxidative Stress
Keywords: PCOS; polycystic ovary syndrome; polycystic ovarian syndrome; alpha lipoic acid; insulin resistance; oxidative stress
MeSH Terms: conditions — Insulin Resistance; Polycystic Ovary Syndrome | interventions — Thioctic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: Alpha Lipoic Acid

SUMMARY:
The study will recruit 40 subjects with Polycystic Ovary Syndrome (PCOS) as defined by the NIH criteria. The subjects will be pre-screened for insulin sensitivity using fasting insulin and glucose levels and oral glucose tolerance test. The 20 most insulin resistant subjects will undergo measurements of in vivo insulin action by hyperinsulinemic, euglycemic clamp. Body composition will be measured by dual-energy X-ray absorptiometry (DEXA). Plasma lipids and markers of oxidative stress will be measured. They will then receive open label controlled release alpha lipoic acid (CRLA) at 800 mg twice daily for 16 weeks. After treatment hyperinsulinemic euglycemic clamps, DEXA, plasma lipids and markers of oxidative stress will be repeated.

Hypotheses: LA will improve insulin sensitivity in PCOS subjects; LA will reduce oxidative stress, testosterone levels and improve cardiovascular risk factors.

DETAILED DESCRIPTION:
Insulin resistance commonly occurs in patients with Polycystic Ovary Syndrome (PCOS) and may be responsible for many of the long term complications of PCOS. Patients with PCOS are at increased risk for developing type 2 diabetes and the metabolic syndrome (hypertension, dyslipidemia and cardiovascular disease). Data suggest that oxidative stress contributes to insulin resistance and thus inhibitors of oxidative stress improve insulin action. Alpha Lipoic Acid (LA) is synthesized in the liver and other tissues and is a key component of several mitochondrial enzyme complexes responsible for oxidative glucose metabolism and cellular energy production. When used pharmacologically, LA functions as a safe and effective antioxidant, recycling vitamins C and E,elevating glutathione levels,and lowering reactive oxygen species. Cell culture studies reveal that LA reverses the effects of oxidative stress and improving insulin action. Preliminary clinical data indicate that antioxidants may improve insulin resistance in PCOS patients. We propose, therefore, to study LA's effects on insulin-stimulated glucose uptake (insulin clamp) in a well characterized population of insulin resistant PCOS patients. Because these patients usually present in the adolescent and teenage years, the development of safe, long-term, treatment strategies are needed.

ELIGIBILITY:
Inclusion Criteria:

* PCOS diagnosis
* 18 years of age or older
* Body Mass Index below 35
* Willing to use any form of contraception for the duration of the study

Exclusion Criteria:

* Diabetes
* Pregnancy
* Liver or heart disease or other health problems
* Taking medications that affect insulin resistance

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2006-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Umesh Masharani, MD, Principal Investigator — University of California, San Francisco; Ira Goldfine, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California at San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Masharani U, Gjerde C, Evans JL, Youngren JF, Goldfine ID. Effects of controlled-release alpha lipoic acid in lean, nondiabetic patients with polycystic ovary syndrome. J Diabetes Sci Technol. 2010 Mar 1;4(2):359-64. doi: 10.1177/193229681000400218. PMID 20307398